CLINICAL TRIAL: NCT03178266
Title: Zip Arthroplasty Patient Satisfaction Evaluation
Acronym: ZAPS
Status: Completed | Type: Observational
Sponsor: ZipLine Medical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 011
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Knee Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Zip Closure Device: Patients will receive the Zip Closure Device for final skin closure after knee arthroplasty.
  Interventions: Device: Knee Arthroplasty
- Metal Staples: Patients will receive Metal Staples for final skin closure after knee arthroplasty.
  Interventions: Device: Knee Arthroplasty

INTERVENTIONS:
Device: Knee Arthroplasty — Standard Knee Arthroplasty will be performed on study subjects. The closure method will be studied at 3 weeks and 6 weeks and patients will be asked about satisfaction with the closure method assigned.

SUMMARY:
This study is a prospective, randomized, single center, study to evaluate Zip Closure Device in subjects undergoing knee arthroplasty. Patients identified as candidates for knee arthroplasty and meet the study selection criteria will be approached and considered for the study. Knee Arthroplasty of 40 subjects will be enrolled where 20 subjects will receive ZipLine and 20 subjects will receive Staples.

DETAILED DESCRIPTION:
Sutures and metal staples are considered standard of care methods for surgical skin closure. The Zip® Surgical Skin Closure device from ZipLine Medical, Inc. (Campbell, CA USA) is a more recent method of skin closure that utilizes skin adhesive and adjustable ratcheting straps to achieve and maintain tension necessary for wound closure and healing. The Zip device was designated Class I, 510(k) Exempt by the US FDA in 2010, and the CE Mark was affixed in 2014.

Limited patient-reported satisfaction data exists for the Zip device as compared to staples and sutures, so this study will attempt to address this need.

The purpose of the study is to evaluate patient satisfaction of closure method used after knee joint arthroplasty. Metal staples and the Zip® Surgical Skin Closure device are approved methods in regular use. Selection of method is generally based on physician preference. This study is to determine what, if any, differences exist in patient satisfaction amongst the two methods

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing primary elective knee arthroplasty.
2. Willing and able to provide informed consent and/or obtain legal guardian authorization
3. Willing and able to comply with the subject-specific requirements outlined in the study protocol

Exclusion Criteria:

1. Patients that do not meet the conditions listed in the wound closure device warnings, precautions, and contraindications (Appendix A)
2. Patients with comorbidities or conditions that the investigator deems to be ineligible for the study
3. Patients without the capacity to give informed consent (e.g., dementia)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Candidates for knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Menkowitz, MD, Principal Investigator — Cheif of Surgery and Orthopaedics
Locations (1):
- Montgomery Orthopaedics Associates, Norristown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zip Closure Device | Metal Staples
Started | 21 | 20
Completed | 21 | 16
Not Completed | 0 | 4
Not completed — Death | 0 | 1
Not completed — Disont. Early | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zip Closure Device | Metal Staples | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (7.13) | 65 (6.96) | 66 (6.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 20 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 17 | 18
  White | 19 | 3 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Patient and Observer Scar Assessment Scale (POSAS)
Description: The subject and investigator will rate commonly described scar characteristics from a patient and observers perspective Subject and Physician will rate overall opinion of scar to normal skin where 1-Normal to 10-Very Different
Time Frame: 6 weeks post knee arthroplasty
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zip Closure Device | Metal Staples
Number analyzed (Participants) | 21 | 16
score on a scale
  Subject Overall Opinion | 2.25 (1.52) | 3.40 (1.96)
  Surgeon Overall Opinion | 1.10 (0.31) | 2.29 (1.10)

2. Secondary Outcome: Patient Satisfaction
Description: Subject Experience and Satisfaction results at 6 weeks post procedure. Subjects are asked of satisfaction with scar appearance on a scale of 1-minimal scar to 5-significant scar
Time Frame: 6 weeks post knee arthroplasty
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zip Closure Device | Metal Staples
Number analyzed (Participants) | 21 | 16
score on a scale | 1.45 (0.76) | 1.94 (0.97)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Zip Closure Device | Metal Staples
All-Cause Mortality (participants affected / at risk) | 0/21 | 1/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/20
Other Adverse Events (participants affected / at risk) | 2/21 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zip Closure Device (N=21) | Metal Staples (N=20)
Death (Cardiac disorders) | 0 (0) | 1 (1) — Cardiac arrest after discharge and before 3 week study visit
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zip Closure Device (N=21) | Metal Staples (N=20)
Blister lateral to distal end of closure (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Serous Drainage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT03178266/Prot_SAP_000.pdf